CLINICAL TRIAL: NCT05262010
Title: A Multicenter Randomized, Blinded, Placebo-controlled Phase III Clinical Trial Evaluating the Protective Efficacy, Safety and Immunogenicity of a 11-valent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) in Chinese Women Aged 9-45 Years
Brief Title: A Phase III Clinical Trial of a 11-valent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) in Chinese Women Aged 9-45 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry); Simoon Record Pharma Information Consulting Co., Ltd. (Industry); Beijing Kantorico Statistical Technology Co., Ltd. (Unknown); Guangxi Center for Disease Control and Prevention (Other Government); Hunan Provincial Center for Disease Control and Prevention (Other); Sichuan Center for Disease Control and Prevention (Other Government); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GXIRB2021-0029-1
Record Dates: First submitted 2022-01-27; First posted 2022-03-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: HPV InfectioN; HPV-Related Carcinoma
Keywords: HPV Infection HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the experiment vaccine
  Interventions: Biological: 11-valent recombinant human papilloma virus vaccine (Hansenula polymorpha)
- placebo (Placebo Comparator): According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: 11-valent recombinant human papilloma virus vaccine (Hansenula polymorpha) — According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the experiment vaccine
  Arms: experiment group
Biological: placebo — According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the placebo
  Arms: placebo

SUMMARY:
A total of 13500 Chinese women aged 18-45 years old were divided into three age groups: 18-26 years old, 27-35 years old, and 35-45 years old. The experimental group and the placebo group were randomly assigned in a ratio of 1:1. All subjects enrolled in the upper arm deltoid muscle were injected with 3 doses of test vaccine or placebo according to the 0, 2, and 6 months immunization program.

ELIGIBILITY:
Inclusion Criteria:

- non-gynecological related

1. *Chinese women with a history of sexual life who are 18-45 years old at the time of enrollment and can provide legal identification;
2. *Axillary body temperature <37.3℃ on the day of enrollment;
3. The subjects themselves have the ability to understand the clinical trial and voluntarily sign the informed consent;
4. Subjects have the ability to read, understand, and fill out research application forms such as diary cards/contact cards, and promise to follow the research requirements participate in follow-up visits;
5. No previous HPV vaccination history, no commercially available HPV vaccine during the study period (about 6 years after enrollment) plan of;
6. The subject has a negative urine pregnancy test on the day before vaccination.

   - Gynecology related
7. *Effective contraception was taken from day 1 of last menstrual cycle to day 0 of the study, and no childbearing within 7 months after enrollment plan.
8. *Before the gynecological visit and within 48 hours before any subsequent visit that includes a gynecological sample collection: asexual life (including same-sex or opposite-sex anal, vaginal or genital contact), unwashed/washed vagina (Except for normal bathing outside the vagina）, no vaginal drugs or preparations are used.

Exclusion Criteria:

First dose exclusion criteria:

(Visits may be rescheduled if the criteria described in the "*" option are met at screening)

- Non-gynecological related

1. * Those with abnormal blood pressure (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg) on physical examination before vaccination;
2. *3 months prior to vaccination or planned to receive any immune globulin or blood products within 7 months of enrollment;
3. *Received any vaccine within 14 days prior to vaccination, or received live vaccine within 28 days;
4. *3 days before vaccination, suffering from acute febrile illness (body temperature ≥38.5℃) or using antipyretic, analgesic and antiallergic drugs (eg: acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
5. History of severe allergies/conditions requiring medical intervention (e.g. Anaphylactic shock, anaphylactic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, local allergic necrosis(Arthus reaction) etc.);
6. Immunocompromised or diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia Blood disease, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammation STD or other autoimmune disease;
7. 1 month before vaccination or plan to receive immunosuppressive therapy within 7 months after enrollment, such as oral administration for more than 2 consecutive weeks Oral or injectable systemic corticosteroid therapy (≥2 mg/kg/day or ≥20 mg/day prednisone or equivalent to prednisone) amount); however, topical medications (such as ointments, eye drops, inhalers, or nasal sprays) are not limited;
8. Previous splenectomy or impaired spleen function;
9. Those with previous or current severe liver, kidney and cardiovascular diseases, complicated diabetes, and malignant tumors;
10. Have a history of epilepsy, convulsions, mental illness or a family history of mental illness;
11. Suffering from thrombocytopenia or any coagulation disorder that can become a contraindication to intramuscular injection;
12. Participate in other clinical studies (drugs, vaccines and medical devices) within 3 months before vaccination or during the planned study period;
13. The investigator believes that the subject has any other factors that are not suitable for participating in the clinical trial (such as: poor compliance or planning Permanent relocation from the area before the study is completed, etc.).

    - Gynecology related
14. *Pregnant, breastfeeding, or within 6 weeks of pregnancy at the time of the first dose of the vaccine;
15. *The subject is in the menstrual period;
16. *Acute lower genital tract infection (such as acute vulvitis/vaginitis/cervicitis, etc.) found by the naked eye during gynecological examination;
17. Previous history of abnormal cervical cancer screening or lesions (including HPV DNA positive, squamous intraepithelial lesion (SIL)or atypical squamous cells of undetermined significance (ASC-US), atypical squamous epithelial cells - excluding high-grade squamous cells Intraepithelial lesions (ASC-H), atypical glandular cells (AGC) or with cervical intraepithelial neoplasia (CIN),Adenocarcinoma in situ (AIS) or cervical cancer, etc.);
18. Past or current anal and genital diseases (such as vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts,vulvar cancer, vaginal cancer and anal cancer, etc.);
19. Previous hysterectomy or pelvic radiation therapy or severe cervical/vaginal dysplasia.

Exclusion criteria for 2nd and 3rd dose vaccination：

If any of the following occurs, the investigator will terminate the subject's vaccination with the investigational vaccine.

* Meet the first dose exclusion criteria 5, 6, 7, 8, 9, 12;
* Any other reasons that, in the judgment of the investigator, warrant discontinuation of the investigational vaccination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 13500 (Estimated)
Dates: Start 2022-06-04 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Person-years incidence of CIN2+ associated with HPV6/11/16/18. | 1 month after 3 doses of vaccine
Person-years incidence of CIN2+ associated with HPV31/33/45/52/58/59/68 | 1 month after 3 doses of vaccine

SECONDARY OUTCOMES:
Person-years incidence of PI12 and PI6 associated with HPV6/11/16/18 types. | 1 month after 3 doses of vaccine
Person-years incidence of PI12 and PI6 associated with HPV31/33/45/52/58 | 1 month after 3 doses of vaccine
Person-years incidence of HPV6/11/16/18/31/33/45/52/58/59/68 types associated with CIN2+, CIN1+, PI12 and PI6 | 1 month after 3 doses of vaccine
Person-years incidence of HPV6/11/16/18/31/33/45/52/58/59/68-associated anogenital and vaginal lesions (including: genital warts, VIN1+, VaIN1+, and AIN1+). | 1 month after 3 doses of vaccine
Person-years incidence of CIN2+, PI12 and PI6 associated with HPV6/11/16/18 | After at least 1 dose of vaccine
Person-years incidence of CIN2+, PI12 and PI6 associated with HPV31/33/45/52/58/59/68 | After at least 1 dose of vaccine
Person-years incidence of CIN2+, CIN1+, PI12 and PI6 associated with HPV6/11/16/18/31/33/45/52/58/59/68 types. | After at least 1 dose of vaccine
Person-years incidence of HPV6/11/16/18/31/33/45/52/58/59/68-associated anogenital and vaginal lesions (including: genital warts, VIN1+, VaIN1+, and AIN1+). | After at least 1 dose of vaccine
AE incidence and severity distribution | The first dose of vaccination to within 1 month after the full vaccination
AE incidence and severity distribution | 0-30 days after each dose vaccination (including 30 minutes, 0-7 days, 8-30 days)
SAE incidence | During the study，an average of 6 year
Number of pregnant | The first dose of vaccination to within 6 months after the full vaccination
Obtain pregnancy outcomes in pregnant subjects( pregnancy event report form) | The first dose of vaccination to within 6 months after the full vaccination
  Previous pregnancy, current pregnancy mode, neonatal information
To evaluate the positive conversion rate of neutralizing antibodies in subjects who completed 3 doses of 11-valent recombinant human papillomavirus vaccine (Hansenula) | 7 (1 month after the first dose), 12, 24, 36, 48, 60 and 72 months after the whole course of vaccination
To evaluate the GMT in subjects who completed 3 doses of 11-valent recombinant human papillomavirus vaccine (Hansenula) | 7 (1 month after the first dose), 12, 24, 36, 48, 60 and 72 months after the whole course of vaccination

OTHER OUTCOMES:
Person-years incidence of PI12 and PI6 associated with HPV59/68 | 1 month after 3 doses of vaccine
Person-years incidence of PI12 and PI6 associated with HPV59/68 | 1 month after 1 doses of vaccine

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Hechi Yizhou District Center for Disease Control and Prevention, Hechi, Guangxi
  - Hezhou Center for Disease Control and Prevention, Hezhou, Guangxi
  - Lianyuan Center for Disease Control and Prevention, Lianyuan, Hunan
  - Qiyang Center for Disease Control and Prevention, Wuxi, Hunan
  - Yongji Center for Disease Control and Prevention, Yongji, Shanxi
  - Yuanqu Center for Disease Control and Prevention, Yuncheng, Shanxi
  - Mianyang Youxian District Center for Disease Control and Prevention, Mianyang, Sichuan
  - Neijiang Shizhong District Center for Disease Control and Prevention, Neijiang, Sichuan

IPD SHARING:
Plan to Share IPD: No